CLINICAL TRIAL: NCT02364401
Title: Comparison of Efficacy Between Impedance Guided and Contact Force Guided Atrial Fibrillation Ablation Using Automated Annotation System
Brief Title: Impedance vs. Contact Force Guided Atrial Fibrillation Ablation Using Automated Annotation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSMCEP_PHS_001
Record Dates: First submitted 2015-01-30; First posted 2015-02-18 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Impedance Guided Ablation Group (Experimental): Impedance guided ablation group performs pulmonary vein(PV) isolation guided by annotation criteria with minimum time of 10 seconds, maximum range of 2 mm, and minimum impedance decrease over 5 Ohms instead of CF parameters. In the impedance guided group, operators are blinded to contact force data during PV isolation.
  Interventions: Device: Ablation
- Contact Forced Guided Ablation Group (Active Comparator): Contact force(CF) guided ablation group performs pulmonary vein (PV) isolation guided by automated annotation criteria with minimum time of 10 seconds, maximum range of 2mm, CF over time of 50% and minimum CF of 10 g.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Catheter ablation for atrial fibrillation
  Other Names: THERMOCOOL® SMARTTOUCH™ catheter

SUMMARY:
The purpose of this study is to compare the efficacy of catheter ablation for atrial fibrillation between contact force-guided and impedance-guided annotation using automated annotation system (Visitag™). Patients who receive atrial fibrillation ablation are randomly assigned in the same number to two groups with impedance guided ablation and contact force guided ablation using contact force sensing catheter (THERMOCOOL® SMARTTOUCH™ catheter, Biosense Webster, Inc., Diamond Bar, CA).

DETAILED DESCRIPTION:
During atrial fibrillation ablation, the location where ablation is conducted is displayed through annotation tags using 3D system to recognize energy delivery is done at the area. However this annotation method was unable to identify how effectively the ablation is done. To remedy this disadvantage, automated annotation system (VisiTag™ module, Biosense Webster, Inc., Diamond Bar, CA) was recently developed to make an automatic annotation when all pre-defined criteria are satisfied. But study on the clinical effects of this system is insufficient.

The purpose of this study is to compare the efficacy of catheter ablation for atrial fibrillation between contact force-guided and impedance-guided annotation using automated annotation system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-valvular atrial fibrillation
* Patients having atrial fibrillation even after receiving continued treatment with at least 1 antiarrhythmic drug for more than 6 weeks
* Patients with tachycardia-bradycardia syndrome associated with atrial fibrillation.
* Patients who can understand the information sheet and consent form on the need and procedure of catheter ablation and submitted them
* Patients who are available of follow-up at least for more than three months after catheter ablation

Exclusion Criteria:

* Patients unsuitable for catheter ablation because the size of left atrium is over 5.5cm
* Patients unsuitable for catheter ablation due to previous history of pulmonary surgery or structural heat disease.
* Patients who cannot receive standard treatments such as anticoagulation therapy which need to be continuously performed prior to radiofrequency catheter ablation
* Patients in the subject group vulnerable to clinical study
* Patients who had undergone a prior catheter ablation for atrial fibrillation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Acute success rate of pulmonary vein isolation obtained after initial circumferential ablation line around pulmonary veins | 6 hours
  Acute success is defined as confirmation of entrance block in all pulmonary veins

SECONDARY OUTCOMES:
Recurrence of any atrial arrhythmias (atrial fibrillation or atrial tachycardia) | 12 months
Procedure time | 6 hours
Ablation time | 6 hours
Average contact force of each ablation lesion | 6 hours
Impedance drop of each ablation lesion | 6 hours
Force time integral of each ablation lesion | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung-Seob Park, MD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea